CLINICAL TRIAL: NCT00118235
Title: Cisplatin, Irinotecan and Bevacizumab (NSC# 704865) for Untreated Extensive Stage Small Cell Lung Cancer: A Phase II Study
Brief Title: Cisplatin, Irinotecan, and Bevacizumab, in Treating Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02815; NCI-2012-02815 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000433341; CALGB-30306 (Other: Cancer and Leukemia Group B); CALGB-30306 (Other: CTEP); U10CA031946 (NIH); P30CA014236 (NIH)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2012-12

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — Cisplatin; Irinotecan; Bevacizumab

ARMS (1):
- Treatment (cisplatin, irinotecan hydrochloride, bevacizumab) (Experimental): Patients receive cisplatin IV over 60 minutes and irinotecan IV over 90 minutes on days 1 and 8. Patients also receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride; Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving cisplatin and irinotecan together with bevacizumab works in treating patients with extensive-stage small cell lung cancer. Drugs used in chemotherapy, such as cisplatin and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of small cell lung cancer by blocking blood flow to the tumor. Giving cisplatin and irinotecan together with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the percentage of patients with extensive stage small cell lung cancer treated with cisplatin, irinotecan and bevacizumab who live longer than 12 months.

SECONDARY OBJECTIVES:

I. To assess the response rate of patients treated with cisplatin, irinotecan and bevacizumab.

II. To evaluate the toxicity and tolerability of the combination of cisplatin, irinotecan and bevacizumab.

III. To determine the association between VEGF/KDR complex expression and VEGF plasma levels and tumor response.

OUTLINE:

Patients receive cisplatin IV over 60 minutes and irinotecan IV over 90 minutes on days 1 and 8. Patients also receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically or cytologically documented small cell carcinoma of the bronchus
* The extensive disease classification for this protocol includes all patients with disease sites not defined as limited stage; limited stage disease category includes patients with disease restricted to one hemithorax with regional lymph node metastases, including hilar, ipsilateral and contralateral mediastinal, and/or ipsilateral supraclavicular nodes; extensive stage patients are defined as those patients with extrathoracic metastases, malignant pleural effusion, bilateral or contralateral supraclavicular adenopathy or contralateral hilar adenopathy
* Measurable or Non-measurable Disease
* No prior chemotherapy or investigational therapy for SCLC
* Radiation therapy must have been completed at least three weeks before initiation of protocol therapy
* No major surgical procedure within 28 days prior to starting treatment and fully recovered
* No minor surgical procedure (mediastinoscopy or core biopsy) within 7 days prior to starting treatment
* ECOG performance status: 0-2
* No "currently active" second malignancy other than non-melanoma skin cancers
* No CNS metastases; patients with a history of CNS metastases will NOT be eligible even if they have completed a course of CNS radiotherapy; all patients will have a screening brain CT or MRI to rule out occult CNS metastases
* No recent history of CVA (within 6 months)
* No serious or non-healing wound ulcer or bone fracture
* Patients with a history of significant bleeding episodes (e.g., hemoptysis, bleeding diathesis, upper or lower GI bleeding) are not eligible; patients with trace blood in the sputum ("blood tinged sputum") are eligible
* No myocardial infarction or significant change in anginal pattern within one year or current congestive heart failure (NYHA Class 2 or higher)
* Patients with a history of hypertension must be well controlled (< 150/90) on a stable regimen of anti-hypertensive therapy
* No HIV-positive patients receiving combination anti-retroviral therapy because of possible pharmacokinetic interactions with the protocol treatment; (patients with immune deficiency are at an increased risk of lethal infections when treated with marrow-suppressive therapy)
* No chronic daily treatment with aspirin (> 325 mg/day) or on non-steroidal antiinflammatory agents known to inhibit platelet function; no treatment with dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix), cilostazol (Pletal), or other antiplatelet agents
* No clinically significant peripheral neuropathy (grade >= 2)
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No treatment with therapeutic anticoagulation; prophylactic anticoagulation for central venous access devices is allowed provided requirements of INR < 1.5 and PTT < 1.2 x ULN are met; caution should be taken in treating patients with low dose heparin or low molecular weight heparin for DVT prophylaxis as there may be an increased bleeding risk with bevacizumab
* No current and/or recent (within 1 month) use of a thrombolytic agent; low dose thrombolytic therapy for maintenance of central venous catheter is allowed
* No clinically significant peripheral arterial disease
* Non-pregnant and non-nursing; the effect of the combination of bevacizumab, cisplatin, and irinotecan on the fetus and infant is unknown
* Granulocytes >= 1,500/μl
* Platelets >= 100,000/μl
* Serum Creatinine =< ULN
* Total Bilirubin < 2.0 mg/dl
* SGOT < 2 x ULN
* INR < 1.5
* PTT < 1.2 x ULN
* Urine protein (dipstick) < 1+

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2004-12; Primary Completion 2007-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Survival time | The time beginning at randomization until death or last known follow-up, assessed up to 4 years
  Described using Kaplan-Meier curves.
Failure-free survival | The time between randomization and the occurrence of disease progression, or death, whichever comes first, assessed up to 4 years
  Described using Kaplan-Meier curves.

SECONDARY OUTCOMES:
Frequency of toxicity, tabulated by the most severe occurrence | Up to 4 years
  Graded using the NCI CTCAE version 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Ready, Principal Investigator — Cancer and Leukemia Group B
Locations (2):
- United States (2):
  - Cancer and Leukemia Group B, Chicago, Illinois
  - Rhode Island Hospital, Providence, Rhode Island